CLINICAL TRIAL: NCT03735381
Title: Efecto de Caminar en La prevención de aparición de Insomnio en el Tercer Trimestre de la gestación. Ensayo de Campo Controlado y Aleatorizado
Brief Title: Walking in Pregnancy and Prevention of Insomnia in Third Trimester Using Pedometers
Acronym: Walking_preg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Carmen Amezcua Prieto, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI-0350-2018
Record Dates: First submitted 2018-11-03; First posted 2018-11-08 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Insomnia
Keywords: Pedometer watch, walking, pregnancy, insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants know they will be selected for either a pedometer group or a not pedometer group. They wil not know if the intervention is minimum (pedometer only) or maximum (pedometer and a goal of 11000 steps/day)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1: pedometer (Active Comparator): Minimum intervention:
  1. Use of pedometer watch from 12 to 32 GW
  2. Recommendations of physical activity
  Interventions: Device: Pedometer watch 'Xiomi mi band2'
- Intervention 2: pedometer+goal+reminds (Experimental): Maximum intervention:
  1. Use of pedometer from 12 to 32 GW
  2. Recommendations of physical activity
  3. Information about get a goal of 11000 steps/day
  4. Reminds the goal every two weeks.
  Interventions: Device: Pedometer watch 'Xiomi mi band2'
- Control: without pedometer (No Intervention): Women receive some recommendations of physical activity during pregnancy. They do not use the pedometer during pregnancy

INTERVENTIONS:
Device: Pedometer watch 'Xiomi mi band2' — 1. They receive information on the use of the pedometer.
  2. Carry the pedometer (Xiaomi Mi Band 2 ™) from 12 to 32GW.
  3. Prescription of benefits of walking in pregnancy:
     * Receive information about the goal of steps / day to be reached: 10,000-11,000 steps / day (Only the intervention 2 group).
     * Receive information on the adequacy of walking with moderate intensity.
  4. They will receive messages on the mobile phone remembering the goal to achieve and a notification that the researching staff will proceed to collect the average count of steps / day of the week prior to 20 and 32 gestation weeks (only for the intervention 2 group).
  Arms: Intervention 1: pedometer; Intervention 2: pedometer+goal+reminds

SUMMARY:
Randomized Control Trial (RCT), were healthy but sedentary women are selected in their first trimester of pregnancy. This RCT has two interventions arms (pedometer plus a goal of 11,000 steps / day and pedometer without goal) and a control group arm, without the use of pedometer. The main objective is to promote physical activity in pregnancy decreasing the prevalence of insomina at their third trimester of pregnancy.

DETAILED DESCRIPTION:
General Objective: To determine the effect of a walking program during pregnancy in the prevention of the appearance of insomnia in the third trimester of pregnancy, in the increase of the quality of sleep and in the improvement of the quality of life throughout pregnancy.

Specific Objectives: Comparison of the interventions group versus the control group; at the beginning, middle and end of the program of the following indicators: 1. Average steps/day; 2. Frequency of insomnia; 3. Hours of night sleep and quality of sleep; 4. Quality of life level.

Methodology: Randomized Control trial in parallel in healthy sedentary pregnant women belonging to the Virgen de las Nieves Hospital in Granada, Spain. At 12 weeks of gestation (GW) they will be invited to participate and randomly assigned to the intervention group I2 (pedometer, with goal of 11,000 steps / day), intervention group I1 (pedometer without goal) and control (without pedometer). Duration of the intervention: 13-32 GW. At 12, 19 and 31GW the average steps/day will be measured in groups I2 and I1. In weeks 13, 20 and 32GW, the following variables will be collected: the Athens Insomnia Scale, the Sleep Quality Index (Pittsburgh), adherence to the Mediterranean Diet (Predimed), physical activity (short IPAQ), quality of life (PSI), the consumption of toxic substances (caffeine, illegal drugs, alcohol and tobacco), the anthropometric variables of pregnant woman.

ELIGIBILITY:
Inclusion Criteria:

* Low risk pregnancies that are attending in the Unit of Obstetrics and Gynecology of the Hospital Materno-Infantil de Granada.
* Sedentary women (<5 days/week of moderate-vigorous physical activity at least >30 min.; equivalent to <7.000 steps/day).
* With mobile phone and e-mail
* Without intellectual deficits or difficulty to understand the language.

Exclusion Criteria:

* Chronic disease: diabetes, high pressure, cardiac or respiratory disease, liver or kidney disease or mobility problems.
* Women with relative or absolute repose.
* Active women (>5 days/week of moderate-vigorous physical activity at least >30 min.; equivalent to >7.000 steps/day).
* Insomnia at beginning of pregnancy or having drugs for sleep problems.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 265 (Estimated)
Dates: Start 2019-06-02 (Actual); Primary Completion 2019-12-15 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Insomnia in third trimester of pregnancy in the three arms with the Insomnia Athens Scale | 32 Gestational Week (GW)
  Insomnia Athens Scale (IAS): An eight-item scale that assesses the quantity and quality of sleep (first five items) and the diurnal repercussion of insomnia (daytime sleepiness, physical and mental functioning and well-being during the day). Each of the items scores from 0 to 3 (affectation of the item from light to severe). The total score ranges from 0 to 24 points, considering insomnia from a score equal to or greater than 6 points (S = 93% and E = 85%) or equal to or greater than 7 points (S = 84% and E = 90%).
Change in mean steps/day after intervention in the arms using pedometer | 19 Gestational Week (GW) and 32 GW
  Pedometer register

SECONDARY OUTCOMES:
Quality of sleep of pregnant women through pregnancy in the three arms measure with the Pittsburgh Questionnaire | 12 (GW), 19 GW and 32 GW
  Pittsburgh Questionnaire (PSQI): it assesses the quality of the individual's sleep during the previous month. It consists of 19 items grouped into seven components: quality, latency, duration, efficiency and sleep disturbances, use of medication for sleep and diurnal dysfunction; each component is scored from 0 to 3, according to a Likert scale in which zero is the absence of the symptom and 3 its maximum presence. This will result in a score that ranges from 0 to 21 points (higher score worse sleep quality): a PSQI score of more than 5 indicates poor sleep quality, with a diagnostic sensitivity of 89.6% and a specificity of 86.5 %.

OTHER OUTCOMES:
Quality of life of women through pregnancy in the three arms measure with the Pregnancy Synpton Inventory | 12 Gestational Week (GW), 19 GW and 32 GW
  Pregnancy Sympton Inventory (PSI): Is a 41-item likert scale developed from a group of experts and focus groups. Registers the range of symptoms that appear in the last month (Likert scale from 0 to 4: never, rarely, sometimes, often) and its impact on quality of life, by affecting the activities of daily life (scale Likert from 0 to 3: it does not limit me, it limits me a little, it limits me a lot). The scale has been adapted to Spanish pregnant women and is reliable (Kappa coefficient range = 0.6-0.9).
Women weight gain in kilograms in the three arms measure with a scale | 12 Gestational Week (GW) and 32 GW
  Women weight gain in kilograms measure with a scale
Weight of the newborn in the three arms collected from the clinical history | Delivery
  Weight of the newborn collected from the clinical history of the women
Gestational week at delibery in the three arms collected from the clinical history of the women | Delivery
  Gestational week at delibery collected from the clinical history of the women

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Amezcua Prieto, Principal Investigator — Universidad de Granada
Locations (1):
- Hospital Virgen de las Nieves, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Benito-Villena R, Cano-Ibanez N, Roman-Galvez RM, Martin-Pelaez S, Khan KS, Martinez-Galiano JM, Mozas-Moreno J, Amezcua-Prieto C. Gestational weight gain and daily life impact of pregnancy symptoms in healthy women: A multivariable analysis. Eur J Obstet Gynecol Reprod Biol. 2024 Dec;303:85-90. doi: 10.1016/j.ejogrb.2024.10.023. Epub 2024 Oct 16. PMID 39432928
- [Derived] Amezcua-Prieto C, Naveiro-Fuentes M, Arco-Jimenez N, Olmedo-Requena R, Barrios-Rodriguez R, Vico-Zuniga I, Manzanares Galan S, Mozas-Moreno J, Jimenez-Moleon JJ, Gallo-Vallejo JL. Walking in pregnancy and prevention of insomnia in third trimester using pedometers: study protocol of Walking_Preg project (WPP). A randomized controlled trial. BMC Pregnancy Childbirth. 2020 Sep 10;20(1):521. doi: 10.1186/s12884-020-03225-y. PMID 32912184